CLINICAL TRIAL: NCT02333448
Title: Diagnostic Value of PCR Genetic Amplification and Mannan Antigenemia Coupled With Antimannan Antibodies in Intensive Care Patients With Suspected Invasive Candidiasis
Brief Title: Evaluate the Performance of Genetic Amplification by Polymerase Chain Reaction (PCR) and the "Mannan Antigenemia and Antimannan Antibodies Couple as a Means of Diagnosis and a Marker of Follow-up in Invasive Candidiasis.
Acronym: EMPIRICAND
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Charles MSD 2014
Record Dates: First submitted 2014-12-05; First posted 2015-01-07 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Invasive Candidiasis; Treatment With Echinocandin
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with suspected invasive candidiasis
  Interventions: Biological: Blood sample taken on the day the treatment is initiated; Biological: Blood sample taken on day 3 after initiation of treatment; Biological: Blood sample taken on day 5 after initiation of; Biological: Blood sample taken on day 7 after initiation of treatment; Biological: Blood sample taken on day 10 after initiation of treatment

INTERVENTIONS:
Biological: Blood sample taken on the day the treatment is initiated
Biological: Blood sample taken on day 3 after initiation of treatment
Biological: Blood sample taken on day 5 after initiation of
Biological: Blood sample taken on day 7 after initiation of treatment
Biological: Blood sample taken on day 10 after initiation of treatment

SUMMARY:
The study consists in taking 4 tubes of blood at different times over a period of 10 days, via a catheter (central venous or arterial catheter) already in place in the usual therapeutic management. These samples will make it possible to measure blood levels of certain markers specific to invasive candidiasis. PCR will be used to quantify fungal load precisely, that is to say the quantity of yeast present in the blood and to monitor this quantity over time.

These samples will be transferred to a specialized unit and stored for a maximum of three years for use at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed about the study
* Patients aged at least 18 years admitted to a medical Intensive Care or general intensive care
* Patients with suspected invasive candidiasis - that is to say:
* Presenting persistent sepsis despite broad-spectrum antibiotherapy for at least 48 hours or targeted antibiotherapy for a documented bacterial infection (sepsis will be defined according to:

  * the usual SIRS criteria, at least 2 of the following 4: temperature > 38°C or < 36°C, tachycardia > 90/min, respiratory rate > 20/min or blood pressure carbon dioxide (PaCO2 ) < 32 mmHg, leukocytosis > 12000/mm3 or < 4000/mm3 or > 10% of immature forms.
  * Persistent hemodynamic instability (impossibility to significantly diminish catecholamine requirement, need for rapid vascular resuscitation > 1000 ml over the previous 24 hours)
* Candida score ≥ 3 with multifocal colonization
* Decision to initiate echinocandin therapy made by the clinician in charge of the patient

Exclusion Criteria:

* Treatment with echinocandin > 1 day in the week preceding inclusion
* Patients not covered by national health insurance
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in a medical Intensive Care Patients with suspected invasive candidiasis
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-06-12 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change from the start of treatment in genomic DNA of Candida sp. by quantitative PCR | At day 1, day 3, day 5, Day 7 and Day 10 after the start of antifungal treatment with echinocandin.

SECONDARY OUTCOMES:
Change from the start of treatment in mannan antigenemia and antimannan antibodies | At day 1, day 5 and day 10 after the start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France